CLINICAL TRIAL: NCT00367107
Title: Autism: Long Term Course and Impact
Brief Title: Autism in Adult Patients and the Effects on Caregivers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Raz Gross, Head, Mental Health Epidemiology, The Gertner Institute for Epidemiology
Other Study IDs: SHEBA-06-4169-RG-CTIL
Record Dates: First submitted 2006-08-21; First posted 2006-08-22 (Estimated); Last update posted 2008-02-06 (Estimated); Status verified 2008-02

CONDITIONS: Autism
Keywords: Autism spectrum disorders; long-term outcomes; caregiver burden; birth cohort; nested case-control study
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Caregiver Burden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background: The number of adults with autism is expected to rise significantly in the near future, due to two main reasons: First, a dramatic increase in the estimates of the prevalence of autism starting in the mid 1980s; Second, the clinical diagnosis of autism was first introduced during the 1950s, and those diagnosed with autism back then are only now entering middle age. Few studies, however, have focused on the outcomes of adult autistic individuals, and very little is known about the course of autism in adulthood and on the familial burden resulting from caring for an autistic adult. We therefore propose to study adult outcomes in autism, and to examine the influence of raising an autistic individual on the parents.

Working hypothesis and aims: The primary objectives of the study are:

1. Determine clinical status and functioning of autistic adults.
2. Study the influence of raising and caring for an individual with autism on the well-being of the parents.

ELIGIBILITY:
Inclusion Criteria:

* Autism or autism spectrum disorder
* Understands the informed consent
* Hebrew Speaker

Exclusion Criteria:

* Severe acute or chronic illness
* Substance abuse
* In control subjects: Autism or autism spectrum disorder in subject or siblings
* In control subjects: participating sibling

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: autisem
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Raz Gros, MD, Principal Investigator — Mental Health Epidemiology & Psychosocial Aspects of Illness, The Gertner Institute for Epidemiology and Health Policy Research
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel